CLINICAL TRIAL: NCT07083622
Title: The Efficacy of Vitamin C Supplementation on Malondialdehid Levels and Disease Activity in Systemic Lupus Erythematosus Patients
Brief Title: Efficacy of Vitamin C Supplementation on Malondialdehid Levels and Disease Activity in SLE Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitas Sriwijaya (Other)
Responsible Party: Principal Investigator, Yuniza, Principal investigator, Division of Allergy Immunology Faculty Member, Department of Internal Medicine, Universitas Sriwijaya/Mohammad Hoesin General Hospital, Universitas Sriwijaya
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: DP0403DXVIII0608ETIK2392024
Record Dates: First submitted 2025-07-01; First posted 2025-07-24 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2025-07

CONDITIONS: Systemic Lupus Erythematosus (SLE)
Keywords: systemic lupus erythematosus; SLE; vitamin c; Malondialdehid; Mex-SLEDAI; disease activity
MeSH Terms: conditions — Lupus Erythematosus, Systemic | interventions — Ascorbic Acid

STUDY DESIGN:
Intervention Model Description: The study was The study was designed as a single-center double-blind randomized controlled clinical trial. Participants were randomized into two groups receiving Vitamin C or placebo
Who Masked: Participant, Care Provider, Investigator
Masking Description: Triple (Participant, Care Provider, Investigator)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vitamin C (Experimental): The patients were given a tablet containing Vitamin C 500 mg twice a day
  Interventions: Dietary Supplement: Vitamin C
- Placebo (Placebo Comparator): The patients were given a placebo capsule with a similar color, shape, size and taste twice a day
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Vitamin C — The patients received vitamin C supplementation
  Arms: Vitamin C
Dietary Supplement: Placebo — Patients received placebo capsules
  Arms: Placebo

SUMMARY:
The study aimed to evaluate the efficacy of vitamin C supplementation compared to placebo towards malondialdehid levels and disease activity with the MEX-SLEDAI score in Systemic Lupus Erythematosus (SLE) patients. The current study was designed as a single-center double-blind randomized controlled clinical trial. The participants were voluntarily recruited ≥ 18 years old SLE patients, with mild to moderate disease activity and did not consumed vitamin C 1 week prior to the trial study. Participants were randomized into two groups receiving vitamin C supplementation, or placebo. Malondialdehid levels and MEX-SLEDAI score were evaluated at the beginning and at the end of the 8 week trial for analysis.

DETAILED DESCRIPTION:
This research is a double blind randomized controlled trial study. The study subjects were 38 patients diagnosed with mild to moderate lupus activity, randomly divided into 2 groups, who received vitamin C supplementation twice daily for 8 weeks and the group that received placebo. Serum malondialdehid levels and the degree of disease activity using MEX-SLEDAI score were measured before and after treatment.

ELIGIBILITY:
Inclusion Criteria

1. All patients diagnosed with mild to moderate systemic lupus erythematosus (SLE).
2. Patients aged over 18 years.
3. Willing to participate in the study by signing an informed consent form.

Exclusion Criteria

1. Pregnant or breastfeeding patients.
2. Patients currently taking vitamin C supplementation within the past 3 days.
3. Patients with other immune-related disorders, either autoimmune or immunocompromised conditions, such as Human Immunodeficiency Virus (HIV) infection.
4. Patients with comorbid diseases.
5. Patients diagnosed with severe SLE or those who have achieved remission.
6. Patients with hemochromatosis.
7. Patients with a history of kidney stones.

Drop-Out Criteria

1. Death before the completion of the study.
2. Patients who stop taking the study medication for more than 3 weeks.
3. Occurrence of severe side effects or worsening of the disease.
4. Hospitalization or symptom worsening during the intervention period.
5. Loss to follow-up.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2024-09-01 (Actual); Primary Completion 2024-11-30 (Actual); Study Completion 2024-11-30 (Actual)

PRIMARY OUTCOMES:
MEX-SLEDAI | From enrollment to the end of the treatment at 8 weeks
  To determine the effectiveness of adding vitamin C compared to placebo towards disease activity in SLE patients, measured with MEX-SLEDAI score
Malondialdehid | From enrollment to the end of the treatment at 8 weeks
  To determine the effectiveness of adding vitamin C compared to placebo towards malondialdehid levels concentration change in SLE patients.

CONTACTS AND LOCATIONS:
Locations (1):
- Mohammad Hoesin General Hospital, Palembang, South Sumatera, Indonesia

REFERENCES:
- [Background] Bojanic, Z. et al. Effects of Methylprednisolone and Vitamin C Therapy on Malondialdehyde Level in Patients With Systemic Lupus Erythematosus. Acta Medica Median. 49, 10-15 (2010).
- [Background] Minami Y, Sasaki T, Arai Y, Kurisu Y, Hisamichi S. Diet and systemic lupus erythematosus: a 4 year prospective study of Japanese patients. J Rheumatol. 2003 Apr;30(4):747-54. PMID 12672194
- [Background] Atik N, Putri Pratiwi S, Hamijoyo L. Correlation between C-reactive Protein with Malondialdehyde in Systemic Lupus Erythematosus Patients. Int J Rheumatol. 2020 Jul 1;2020:8078412. doi: 10.1155/2020/8078412. eCollection 2020. PMID 32695177